CLINICAL TRIAL: NCT04643171
Title: Markers of Oxidative Stress in Response to Electroacupuncture Against Aerobic Physical Activity in Diabetic Patients
Brief Title: Oxidative Stress in Response to Electroacupuncture Against Physical Activity in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002898
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): 30 patients will receive 30 minutes of high intensity interval training on elliptical trainer, 5 times per week, for 12 week
  Interventions: Device: high intensity elliptical training
- group of electroacupuncture (Active Comparator): 30 patients will receive 30 minutes of electroacupuncture on bilateral PC 4 and PC 6, 5 times per week, for 12 week
  Interventions: Device: electrocaupuncture

INTERVENTIONS:
Device: high intensity elliptical training — 30 patients will receive 30 minutes of high intensity interval training on elliptical trainer, 5 times per week, for 12 week
  Arms: Exercised group
Device: electrocaupuncture — 30 patients will receive 30 minutes of electroacupuncture on bilateral PC 4 and PC 6 for 5 times per week, for 12 week
  Arms: group of electroacupuncture

SUMMARY:
OS is an important pathogenetic mechanism for the development of T2DM and its complications.

Oxidative stress is an imbalance of the generation of free radicals or known as reactive oxygen species (ROS) and reactive nitrogen species [RNS]) and their neutralization by the antioxidant mechanisms.

Increased levels of ROS and RNS lead to damage of lipids, proteins, and DNA, ultimately causing the destruction of the islet cells of pancreas through apoptosis . Elliptical trainer device is a relatively new modality of exercise and is advertised to be superior to a treadmill because of the low joint impact and the more reasonable costs of an elliptical trainer compared to a treadmill . Additional quantative research is needed to further evaluate the effectiveness of elliptical trainers and the physiological and perceptual responses to the machine Electroacupuncture (EA) is a treatment form of traditional acupuncture in which small electrical currents are passed through needles inserted into the subject's skin using EA stimulator. It seems to have more acceptable results and effects on many important clinical applications and medical research sets .

DETAILED DESCRIPTION:
60 diabetic patients will be randomly divided to electroacupucture group (30 patients) and high intensity elliptical training (30 patients). the treatment will be done for 5 sessions per week for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic elderly
* Body mass index less than 30 kg/m2.
* Fasting blood more than 126 mg/dl

Exclusion Criteria:

* cardiac patients
* renal patients
* respiratory patients
* liver patients
* patients who received any complementary therapies within 3 past months

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 60 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
superoxide dismutase | It will be measured after 12 weeks
  marker of anti-oxidative stress

SECONDARY OUTCOMES:
nitric oxide | It will be measured after 12 weeks
  will be measured in plasma
lipid hydroperoxidase | It will be measured after 12-week training
  will be measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt